CLINICAL TRIAL: NCT07403981
Title: Advocacy, Partnership, Outreach, and Yielding Optimized Care for Oncology Patients (APOYO): A Community Health Worker Intervention for Latinx Colorectal Cancer Patients
Brief Title: Advocacy, Partnership, Outreach, and Yielding Optimized Care for Oncology Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-82643
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Worker (CHW)/Patient Navigator (Intervention Group) (Experimental): Participants randomized to the intervention group will be assigned a CHW/P who will provide support for up to 6 months after randomization. CHW/Ps will attend the initial oncology visit when possible, review and explain the treatment plan, assist with scheduling and logistics (e.g., transportation, language services), complete a social needs assessment, connect patients to social support services, and offer peer support connections. CHW/Ps will maintain regular contact with patients, at least every other week for the first 3 months, and be available by phone as needed for an additional 3 months. They will also alert the clinical team if the patient expresses unresolved concerns or questions.
  Interventions: Behavioral: CHW/P Navigator Support
- Usual Care plus Social Services Resource List (Control Group) (Active Comparator): Participants in the control group will receive a printed or digital list of local social service resources, including websites and phone numbers, but will not receive CHW/P support or navigation services.
  Interventions: Other: Social Services Resource List

INTERVENTIONS:
Behavioral: CHW/P Navigator Support — A Community Health Worker/Patient Navigator provides care coordination, social needs assessment, assistance accessing services, logistical support, and ongoing contact for up to 6 months following randomization.
  Arms: Community Health Worker (CHW)/Patient Navigator (Intervention Group)
Other: Social Services Resource List — Participants receive a printed or digital list of local social service resources, including websites and phone numbers for enrollment and access to services.
  Arms: Usual Care plus Social Services Resource List (Control Group)

SUMMARY:
This study is a pilot feasibility randomized trial involving newly diagnosed colorectal cancer (CRC) patients who identify as Latinx. The study aims to leverage existing academic-community partnerships in Santa Clara County to develop and evaluate a multi-level community health worker/promotora (CHW/P) navigator intervention. If found effective, APOYO has the potential to affect clinical outcomes for Latinx colorectal cancer patients both directly and indirectly, including improving health-related quality of life, health care utilization, and reducing social needs.

ELIGIBILITY:
Inclusion Criteria:

1. New diagnosis of colon or rectal cancer in the last 30 days
2. Identify as Latinx/Hispanic/Latino
3. Aged 18 years or older
4. Reside in and planning to receive care in Santa Clara County
5. Ability to understand and the willingness to provide written informed consent

Exclusion Criteria:

1. Unable to speak and understand either Spanish or English
2. Any concurrent malignancy other than nonmelanoma skin cancer or carcinoma in situ of the cervix. Patients with any previous malignancy without evidence of disease for >3 years will be allowed to enter the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Score (EORTC QLQ-C30) | Baseline to 6 months after randomization
  Quality of life measured using the EORTC QLQ-C30 questionnaire, comparing participants randomized to CHW/P navigator support versus usual care with social services resource list.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron J Dawes, MD, PhD, FACS, FASCRS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States